CLINICAL TRIAL: NCT04672395
Title: A Double-blind, Randomized, Controlled, Phase 2/3 Study to Evaluate the Efficacy, Immunogenicity, and Safety of CpG 1018/Alum-Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Subunit Vaccine (SCB-2019) for the Prevention of SARS-CoV-2- Mediated COVID-19 in Participants Aged 12 Years and Older
Brief Title: A Controlled Phase 2/3 Study of Adjuvanted Recombinant SARS-CoV-2 Trimeric S-protein Vaccine (SCB-2019) for the Prevention of COVID-19
Acronym: SCB-2019
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Clover Biopharmaceuticals AUS Pty (Industry)
Collaborators: Coalition for Epidemic Preparedness Innovations (Other); International Vaccine Institute (Other)
Responsible Party: Sponsor
Organization: Clover Biopharmaceuticals, Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLO-SCB-2019-003
Record Dates: First submitted 2020-12-16; First posted 2020-12-17 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Sodium Chloride; SCB-2019 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Each subject will receive 2 doses of their assigned treatment on Days 1 and 22. Booster dose will be given at least 4 months after the second dose (Day 1A for booster dose). The treatment will be administered IM in the deltoid region of the upper non-dominant arm
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): CpG 1018/Alum-adjuvanted SCB-2019 vaccine
  Interventions: Biological: CpG 1018/Alum-adjuvanted SCB-2019 vaccine
- Group 2 (Placebo Comparator): Placebo Comparator: 0.9% Saline
  Interventions: Biological: Placebo; 0.9% saline
- Booster dose of SCB-2019 (Experimental): Adult SCB-2019 recipients will receive 1 dose of SCB-2019 at least 4 months after the second dose
  Interventions: Biological: SCB-2019 vaccine
- Vaccination of placebo recipients with SCB-2019 (Placebo Comparator): Placebo participants will be offered two doses of SCB-2019 vaccine
  Interventions: Biological: SCB-2019 vaccine for Placebo

INTERVENTIONS:
Biological: CpG 1018/Alum-adjuvanted SCB-2019 vaccine — Group 1: Participants will receive 1 intramuscular (IM) injection of 30 microgram (ug) SCB-2019 with CpG1018/Alum adjuvant on Day 1 and on Day 22
  Arms: Group 1
Biological: Placebo; 0.9% saline — Group 2: Participants will receive 1 IM injection of SCB-2019-matching placebo on Day 1 and on Day 22
  Arms: Group 2
Biological: SCB-2019 vaccine — Participants will receive 1 IM injection of 30 microgram (ug) SCB-2019 with CpG 1018/alum adjuvant
  Arms: Booster dose of SCB-2019
Biological: SCB-2019 vaccine for Placebo — Participants will receive 2 IM injection of 30 microgram (ug) SCB-2019 with CpG 1018/alum adjuvant, 21 days apart
  Arms: Vaccination of placebo recipients with SCB-2019

SUMMARY:
The purpose of this double-blind, randomized, controlled study is to evaluate the efficacy, immunogenicity, reactogenicity and safety of an adjuvanted recombinant severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) trimeric spike (S)-protein subunit vaccine (SCB-2019) for the prevention of SARS-CoV-2-mediated COVID-19 in Participants Aged 12 Years and Older.

DETAILED DESCRIPTION:
This study will assess the efficacy against COVID-19, immunogenicity, reactogenicity, and safety of CpG 1018/Alum-adjuvated SCB-2019 vaccine. The COVID-19 pandemic has resulted in high morbidity and mortality, caused major disruption to healthcare systems, and has had significant socioeconomic impacts. Currently, only limited treatment options are available against COVID-19 and accelerated vaccine development is urgently needed. Several COVID-19 vaccines were recently authorized in some countries, but the global supply is insufficient for pandemic control. Additional safe and effective vaccines for COVID-19 prevention would have significant public health impact.

Placebo recipients will be offered two doses of SCB-2019 vaccine at defined points as part of the study.

Adults participants who received SCB-2019 vaccine, will be given a third dose of the SCB-2019 vaccine at least 4 months after the second dose to assess the safety and efficacy of a booster (third) dose.

ELIGIBILITY:
Inclusion Criteria:

1. Male or females ≥12 years of age, inclusive*.
2. Participants who are willing and able to comply with study requirements, including all scheduled visits, vaccinations, laboratory tests, the electronic completion of the COVID-19 ePRO and other study procedures.
3. Healthy adult or adolescent subjects or adult or adolescent subjects with pre-existing medical conditions who are in stable condition. A stable medical condition is defined as disease not requiring significant change in therapy or hospitalization for worsening disease during the 3 months before enrollment.

   *Note: The first 200 individuals enrolled in the Phase 2 part of the study should be healthy subjects 18 to 64 years or age without comorbidities associated with a high risk of severe COVID-19
4. Female subjects who are WOCBP are eligible to participate in the study if not pregnant, not breastfeeding, and at least 1 of the following criteria apply:

   * WOCBP must have a negative urine pregnancy test prior to each vaccination. A confirmatory serum pregnancy test may be conducted at the investigator's discretion.
   * They must be using a highly effective licensed method of birth control for 30 days prior to the first vaccination and must agree to continue such precautions during the study until 90 days after the second vaccination.
5. Male subjects must agree to employ acceptable contraception from the day of first dose of the study vaccine/placebo until 6 months after the last dose of the study vaccine/placebo and also refrain from donating sperm during this period.
6. Individuals (or their legally acceptable representative based on local regulations) willing and able to give an informed consent, prior to screening. For adolescent subjects: informed assent signed by adolescents and informed consent signed by the parent(s) or legally acceptable representative(s) as per local requirements.
7. Applicable for HIV-positive individuals only if:

They are medically stable at screening, as determined by the investigator, and free of opportunistic infections in the 1 year prior to first study vaccination, and They have an HIV-1 viral load <1000 copies/mL within 45 days of randomization in the study, and They are receiving highly active antiretroviral therapy (HAART) for at least 3 months before screening. Changes in antiretroviral dosage within 3 months of entering the study are allowed, as are exchanges in pharmacological formulations.

Exclusion Criteria:

1. Individuals with laboratory-confirmed SARS-CoV-2 infection (e.g., a positive RT-PCR* or Rapid COVID-19 Antigen test) at screening or within 14 days prior to enrollment.
2. Individuals with behavioral or cognitive impairment (including drug and alcohol abuse) in the opinion of the investigator.
3. Individuals with any progressive or severe neurologic disorder, seizure disorder, or history of Guillian-Barré syndrome.
4. Individuals who receive treatment with immunosuppressive therapy, including cytotoxic agents or systemic corticosteroids, e.g., for cancer or an autoimmune disease, or planned receipt during the study period.
5. Individuals who are pregnant, or breastfeeding, or planning to become pregnant during the study period.
6. Individuals who have a history of severe adverse reaction associated with a vaccine or severe allergic reaction (e.g., anaphylaxis) to any component of the study vaccine (SCB-2019, CpG1018 Adjuvant and Aluminum hydroxide components).
7. Individuals who have a history of malignancy within 1 year before screening (exceptions are squamous and basal cell carcinomas of the skin and carcinoma in situ of the cervix which have been cured, or other malignancies with minimal risk of recurrence).
8. Individuals who have received any other investigational product within 30 days prior to Day 1 or intent to participate in another clinical study at any time during the conduct of this study.
9. Individuals who have received previous vaccination with any coronavirus vaccine.
10. Individuals who have received any other licensed vaccines within 14 days prior to enrollment in this study or who are planning to receive any vaccine up to 14 days after the second vaccination.
11. Individuals with known bleeding disorder that would, in the opinion of the investigator, contraindicate intramuscular injection.
12. Individuals who received any blood/plasma products or immunoglobulins within 60 days prior to Day 1 or plan to receive it during the study period.
13. Individuals with any condition that, in the opinion of the investigator, may increase the risk of study participation or interfere with the assessment of the primary study objectives.
14. Individuals with fever >37.8°C (irrespective of method), or any acute illness at baseline (Day 1) or within 3 days of randomization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 31454 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2023-04-23 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a First Occurrence of COVID-19 of Any Severity Starting 14 Days after Second Dose of SCB-2019 | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to Day 8 (7 days after first dose) and up to Day 29 (7 days after second dose)
Number of Participants with Unsolicited AEs | Up to Day 43 (21 days after each dose)
Number of Participants with Serious Adverse Events (SAEs), or Medically Attended AEs (MAAEs), or AEs Leading to Early Termination, or Adverse Events of Special Interest (AESIs) | Up to Day 389 (1 year after second dose)
Non-inferiority of the neutralizing titers after third dose compared to the neutralizing titers after second dose | 14 days after third dose
Non-inferiority of the neutralising titers in adolescents versus young adults. | 14 days after second dose

SECONDARY OUTCOMES:
Number of Participants with a First Occurrence of Moderate-to-Severe COVID-19 Starting 14 Days after Second Dose of SCB-2019 | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with First Occurrence of Any Laboratory-Confirmed SARS-CoV-2 infection Starting 14 Days after Second Dose of SCB-2019 or Placebo | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with a First Occurrence of Severe COVID-19 Starting 14 Days after Second Dose of SCB-2019 or Placebo | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with First Occurrence of Any Laboratory-Confirmed Asymptomatic SARS-CoV-2 infection Starting 14 Days after Second Dose of SCB-2019 or Placebo | Day 36 up to Day 389 (1 year after second dose)
Burden of Disease Score of COVID-19 or SARS-CoV-2 Infection Cases Starting 14 Days after Second Dose of SCB-2019 or Placebo | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with a First Occurrence of COVID-19 of Any Severity, Associated with Hospitalization, Starting 14 Days after Second Dose of SCB-2019 or Placebo | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with a First Occurrence of COVID-19 Starting 14 days after Second Dose of SCB-2019 or Placebo, regardless of evidence of prior SARS-CoV-2 Infection | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with a First Occurrence of COVID-19 Starting 14 days after Second Dose of SCB-2019 or Placebo, regardless of risk of severe COVID-19 | Day 36 up to Day 389 (1 year after second dose)
Number of Participants with a First Occurrence of COVID-19 Starting 14 days after First Dose of SCB-2019 or Placebo | Day 15 up to Day 22
Number of Participants with a First Occurrence of COVID-19 of Any Severity caused by SARS-CoV-2 variants of concern starting 14 days after Second Dose | Day 36 up to Day 389 (1 year after second dose)
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific Neutralizing Antibody (nAb) | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Specific nAb | Day 1, Day 22, Day 35, Day 205, and Day 389
Number of Participants with Seroconversion for SARS-CoV-2 Specific nAb | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Titer (GMT) of SARS-CoV-2 antibodies competing for binding of S protein to the human ACE2 receptor | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 antibodies competing for binding of S protein to the human ACE2 receptor | Day 1, Day 22, Day 35, Day 205, and Day 389
Number of Participants with Seroconversion for of SARS-CoV-2 antibodies competing for binding of S protein to the human ACE2 receptor | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Titer (GMT) of SCB-2019 binding antibody | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Fold Rise (GMFR) of SCB-2019 binding antibody | Day 1, Day 22, Day 35, Day 205, and Day 389
Number of Participants with Seroconversion for SCB-2019 binding antibody | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Titer (GMT) of Trimer-Tag binding antibody | Day 1, Day 22, Day 35, Day 205, and Day 389
Geometric Mean Fold Rise (GMFR) of Trimer-Tag binding antibody | Day 1, Day 22, Day 35, Day 205, and Day 389
Number of Participants with Solicited Local and Systemic Adverse Reactions (ARs) | Up to 7 days after booster dose
Number of Participants with Unsolicited AEs | Up to 21 days after booster dose
Number of Participants with Serious Adverse Events (SAEs), or Medically Attended AEs (MAAEs), or AEs Leading to Early Termination, or Adverse Events of Special Interest (AESIs) | Up to 6 months after booster dose
Geometric Mean Titer (GMT) of SARS-CoV-2 Specific nAb | Day 1A, Day 15A (15 days after booster), and Day 389A (6 months after booster)
Geometric Mean Fold Rise (GMFR) of SARS-CoV-2 Specific nAb | Day 1A, Day 15A (15 days after booster), and Day 389A (6 months after booster)
Number of Participants with Seroconversion for SARS-CoV-2 Specific nAb | Day 1A, Day 15A (15 days after booster), and Day 389A (6 months after booster)
Geometric Mean Titer (GMT) of SCB-2019 binding antibody | Day 1A, Day 15A (15 days after booster), and Day 389A (6 months after booster)
Geometric Mean Fold Rise (GMFR) of SCB-2019 binding antibody | Day 1A, Day 15A (15 days after booster), and Day 389A (6 months after booster)
Number of Participants with Seroconversion for SCB-2019 binding antibody | Day 1A, Day 15A (15 days after booster), and Day 389A (6 months after booster)

CONTACTS AND LOCATIONS:
Overall Officials: Igor Smolenov, MD, PhD, Study Chair — Clover Biopharmaceuticals AUS Pty
Locations (31):
- Belgium (3):
  - Anima, Alken
  - Hôspital Erasme, Brussels
  - Private Practice RESPISOM Namur, Namur
- Brazil (5):
  - Instituto D'OR de Pesquisa e Ensino, Rio de Janeiro, Rio Do Janeiro
  - Instituto Atena de Pesquisa Clinica, Natal, Rio Grande do Norte
  - CPCLIN - Centro de Pesquisas Clínicas de Natal, Natal, Rio Grande do Norte
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital da Universidade Federal de Santa Maria CEP/UFSM, Santa Maria, Rio Grande do Sul
- Colombia (9):
  - Centro de Atención e investigación Médica S.A.S, CAIMED S.A.S - sede, Acacias, Acacías
  - Centro de Atención e investigación Médica S.A.S, CAIMED S.A.S - sede Aguazul, Aguazul
  - Clínica de la Costa Ltda, Barranquilla
  - Fundación Hospital Universitario del Norte, Barranquilla
  - Centro de Atención e investigación Médica S.A.S, CAIMED S.A.S - sede, Bogotá D.C., Bogotá
  - Policlinico Social del Norte, Bogotá
  - Centro de Estudios en Infectología Pediátrica S.A.S. - CEIP S.A.S., Cali
  - IPS Médicos Internistas de Caldas SAS, Manizales
  - Centro de Atención e investigación Médica S.A.S, CAIMED S.A.S - sede, Yopal, Yopal
- Philippines (10):
  - De La Salle Medical and Health Sciences Institute, Dasmariñas, Cavite
  - Asian Hospital and Medical Center, City of Muntinlupa
  - St. Luke's Medical Center, City of Taguig
  - Las Pinas Doctors Hospital, Las Piñas
  - Tropical Disease Foundation, Makati
  - Manila Doctors Hospital, Manila
  - University of the Philippines Manila - Philippine General Hospital, Pasay
  - UERM Memorial Medical Center, Quezon City
  - University of the East Ramon Magsaysay Memorial Medical Center, Quezon City
  - FEU-NRMF Medical Center, Quezon City
- South Africa (4):
  - Wits Clinical Research, Johannesburg, Gauteng
  - DJW Research, Krugersdorp, Gauteng
  - Soweto Clinical Trials Centre, Soweto, Gauteng
  - Dr JM Engelbrecht Trial Site, Somerset West, Western Cape

REFERENCES:
- [Background] Liu H, Su D, Zhang J, Ge S, Li Y, Wang F, Gravel M, Roulston A, Song Q, Xu W, Liang JG, Shore G, Wang X, Liang P. Improvement of Pharmacokinetic Profile of TRAIL via Trimer-Tag Enhances its Antitumor Activity in vivo. Sci Rep. 2017 Aug 21;7(1):8953. doi: 10.1038/s41598-017-09518-1. PMID 28827692
- [Background] Ruggeberg JU, Gold MS, Bayas JM, Blum MD, Bonhoeffer J, Friedlander S, de Souza Brito G, Heininger U, Imoukhuede B, Khamesipour A, Erlewyn-Lajeunesse M, Martin S, Makela M, Nell P, Pool V, Simpson N; Brighton Collaboration Anaphylaxis Working Group. Anaphylaxis: case definition and guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2007 Aug 1;25(31):5675-84. doi: 10.1016/j.vaccine.2007.02.064. Epub 2007 Mar 12. No abstract available. PMID 17448577
- [Background] Rhodes SJ, Knight GM, Kirschner DE, White RG, Evans TG. Dose finding for new vaccines: The role for immunostimulation/immunodynamic modelling. J Theor Biol. 2019 Mar 21;465:51-55. doi: 10.1016/j.jtbi.2019.01.017. Epub 2019 Jan 10. PMID 30639297
- [Background] Food and Drug Administration letter. Device: BinaxNOW COVID-19 Ag Card. 26 August 2020. https://www.fda.gov/media/141567/download. Accessed on 15 September 2020.
- [Background] Amai M, Nojima M, Yuki Y, Kiyono H, Nagamura F. A review of criteria strictness in "Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials". Vaccine. 2023 Aug 31;41(38):5622-5629. doi: 10.1016/j.vaccine.2023.07.072. Epub 2023 Aug 1. PMID 37532612
- [Background] Safety Platform for Emergency vACcines (SPEAC). D2.3 Priority List of Adverse Events of Special Interest: COVID-19. V1.1 Date 05 March 2020. https://media.tghn.org/articles/COVID-19_AESIs_SPEAC_V1.1_5Mar2020.pdf. Accessed on 15 September 2020.
- [Background] Chan ISF, Bohidar NR (1998) Exact power and sample size for vaccine efficacy studies, Communications in Statistics - Theory and Methods 1998;27(6):1305-22.
- [Background] Maurer W, Bretz F. Multiple testing in group sequential trials using graphical approaches. Stat Biopharm Res 2013;5(4):311-20.
- [Derived] Aziz AB, Sugimoto JD, Hong SL, You YA, Bravo L, Roa C Jr, Borja-Tabora C, Montellano MEB, Carlos J, de Los Reyes MRA, Alberto ER, Salvani-Bautista M, Kim HY, Njau I, Clemens R, Marks F, Tadesse BT. Indirect effectiveness of a novel SARS-COV-2 vaccine (SCB-2019) in unvaccinated household contacts in the Philippines: A cluster randomised analysis. J Infect. 2024 Oct;89(4):106260. doi: 10.1016/j.jinf.2024.106260. Epub 2024 Aug 30. PMID 39218309
- [Derived] Lopez P, Bravo L, Buntinx E, Borja-Tabora C, Velasquez H, Rodriquez EJ, Rodriguez CA, Carlos J, Montellano MEB, Alberto ER, Salvani-Bautista M, Huang Y, Hu B, Li P, Han HH, Baccarini C, Smolenov I. Safety and immunogenicity of SCB-2019, an adjuvanted, recombinant SARS-CoV-2 trimeric S-protein subunit COVID-19 vaccine in healthy 12-17 year-old adolescents. Hum Vaccin Immunother. 2023 Dec 31;19(1):2206359. doi: 10.1080/21645515.2023.2206359. Epub 2023 May 25. PMID 37226504
- [Derived] Hosain R, Aquino P, Baccarini C, Smolenov I, Li P, Qin H, Verhoeven C, Hu B, Huang Y, Rubio P; SPECTRA Study Group. Six-month safety follow-up of an adjuvanted SARS-CoV-2 trimeric S-protein subunit vaccine (SCB-2019) in adults: A phase 2/3, double-blind, randomized study. Vaccine. 2023 Mar 24;41(13):2253-2260. doi: 10.1016/j.vaccine.2023.02.018. Epub 2023 Feb 10. PMID 36868877
- [Derived] Buntinx E, Brochado L, Borja-Tabora C, Yu CY, Alberto ER, Montellano MEB, Carlos JC, Toloza LB, Hites M, Siber G, Clemens R, Ambrosino D, Qin H, Chen HL, Han HH, Hu B, Li P, Baccarini C, Smolenov I. Immunogenicity of an adjuvanted SARS-CoV-2 trimeric S-protein subunit vaccine (SCB-2019) in SARS-CoV-2-naive and exposed individuals in a phase 2/3, double-blind, randomized study. Vaccine. 2023 Mar 10;41(11):1875-1884. doi: 10.1016/j.vaccine.2023.02.017. Epub 2023 Feb 9. PMID 36781334
- [Derived] Tadesse BT, Bravo L, Marks F, Aziz AB, You YA, Sugimoto J, Li P, Garcia J, Rockhold F, Clemens R; Household Contact Study Group. Impact of Vaccination With the SCB-2019 Coronavirus Disease 2019 Vaccine on Transmission of Severe Acute Respiratory Syndrome Coronavirus 2 Infection: A Household Contact Study in the Philippines. Clin Infect Dis. 2023 Apr 3;76(7):1180-1187. doi: 10.1093/cid/ciac914. PMID 36433685
- [Derived] Bravo L, Smolenov I, Han HH, Li P, Hosain R, Rockhold F, Clemens SAC, Roa C Jr, Borja-Tabora C, Quinsaat A, Lopez P, Lopez-Medina E, Brochado L, Hernandez EA, Reynales H, Medina T, Velasquez H, Toloza LB, Rodriguez EJ, de Salazar DIM, Rodriguez CA, Sprinz E, Cerbino-Neto J, Luz KG, Schwarzbold AV, Paiva MS, Carlos J, Montellano MEB, de Los Reyes MRA, Yu CY, Alberto ER, Panaligan MM, Salvani-Bautista M, Buntinx E, Hites M, Martinot JB, Bhorat QE, Badat A, Baccarini C, Hu B, Jurgens J, Engelbrecht J, Ambrosino D, Richmond P, Siber G, Liang J, Clemens R. Efficacy of the adjuvanted subunit protein COVID-19 vaccine, SCB-2019: a phase 2 and 3 multicentre, double-blind, randomised, placebo-controlled trial. Lancet. 2022 Jan 29;399(10323):461-472. doi: 10.1016/S0140-6736(22)00055-1. Epub 2022 Jan 20. PMID 35065705